CLINICAL TRIAL: NCT01306149
Title: Natural History of Biochemical Parameters of Mineral Metabolism and Protein-bound Uremic Retention Molecules in Incident Peritoneal Dialysis Patients: a Longitudinal Observational Study
Brief Title: Natural History of Mineral Metabolism Parameters and Protein-bound Toxins in Incident Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Björn Meijers, Dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: FWO01-03-21
Record Dates: First submitted 2011-02-23; First posted 2011-03-01 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Complication of Peritoneal Dialysis
Keywords: biochemical parameters; mineral metabolism; protein-bound uremic retention solutes; incident PD patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, urine and dialysate
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of this study are

1. To evaluate the natural history of plasma concentrations and renal and peritoneal clearances of small water-soluble uremic retention molecules (URM), 'middle molecules', and protein bound URM in incident peritoneal dialysis (PD) patients.
2. To evaluate the natural history and determinants of the generation rate of URM originating from bacterial protein fermentation in PD patients.
3. To evaluate the natural history of biochemical parameters of mineral metabolism in incident PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Incident PD patients, defined as patients who started on PD as first renal replacement therapy less than 8 weeks before inclusion
* written informed consent
* age > 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident peritoneal dialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2002-07 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
natural history of clearances and serum parameters of mineral metabolism and protein-bound toxins | 15 years
  To evaluate the natural history of plasma concentrations and renal and peritoneal clearances of small water-soluble uremic retention molecules (URM), 'middle molecules, and protein bound URM in incident peritoneal dialysis (PD) patients.

SECONDARY OUTCOMES:
determinants of generation rate of uremic retention solutes | 15 years on average
  To evaluate the natural history and determinants of the generation rate of URM originating from bacterial protein fermentation in PD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD,PhD, Principal Investigator — University Hospital, Leuven, Belgium
Locations (1):
- University Hospital, Leuven, Vlaams-Brabant, Belgium